CLINICAL TRIAL: NCT03320863
Title: A Multicenter Randomized Controlled Clinical Trial Evaluating the Effectiveness of a Novel Form of Non-Invasive Neuromodulation for Treatment of Chronic Low Back Pain
Brief Title: The Enso Study for Chronic Low Back Pain
Acronym: EPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thimble Bioelectronics, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol 17-01
Record Dates: First submitted 2017-10-17; First posted 2017-10-25 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, sham controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Devices are assigned per the randomization schedule, with the sham device identical to the active device in every way except that no neuromodulation is delivered. The neuromodulation that the active device delivers can be done in a way that causes no sensation, so subjects are not unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active or Enso Group (Active Comparator): Active Enso device use for one month, at least one hour daily, including coaching via a smartphone app and coaching phone calls regarding device usage.
  Interventions: Device: Enso device
- Sham Group (No Intervention): Sham device use for one month, at least one hour daily, including coaching via a smartphone app and coaching phone calls regarding device usage.

INTERVENTIONS:
Device: Enso device — An active Enso device that delivers neuromodulation therapy.
  Arms: Active or Enso Group

SUMMARY:
Enso is a portable device for the treatment of chronic and acute types of musculoskeletal pain. This study is being designed as a double-blinded, sham-controlled randomized clinical trial.

DETAILED DESCRIPTION:
Fifty subjects will be selected based on the inclusion criteria and then randomized to either the intervention group or the sham control group. Each subject will be randomly fitted with an Enso or a sham device and will be instructed to self-administer treatment daily for one hour or more per day for four weeks in both cohorts. Throughout the duration of the study, data will be recorded via a smartphone application regarding treatment usage and intensity, pain levels, the subject's impression of any changes in their functionality, and their opioid and non-opioid medication intake. Medication usage will also be tracked through the use of CURES 2.0 information and pill counts at specified study visits. Additional functional testing will be conducted at each study visit.

At the 4 week visit, the study blind will be broken, and subjects who were randomized to the sham group will be given the opportunity to cross over for an additional week in the study, using the active device.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical (myofascial), axial back pain (focused around the spine)
2. 6/10 or greater level of pain
3. Functionally debilitated by their pain (e.g., difficulty walking)
4. Minimal radicular symptoms with no effect on functionality, medication, quality of life
5. Expressed desire to stop taking pain medications
6. Expressed desire to improve disability
7. 80% or greater of disability is due to pain in the low back (as opposed to other body areas)
8. Experiencing chronic pain for at least 6 months
9. Interested in being active, improving their functionality
10. Comfortable with using technology in daily life
11. Subject able to understand and grant informed consent
12. Documented adherence with clinic follow up visits per medical records
13. Has an email account
14. Above 18 years old

Exclusion Criteria:

1. Patients that do not own or have access to a smartphone
2. Has spinal instability, joint instability, or grade 2 or greater spondylolisthesis with instability
3. Primary symptoms due to spinal stenosis
4. Source of back pain related to an acute nerve impingement
5. Diagnosis of cancer/malignant tumors in the last 5 years
6. Source of back pain is an infection
7. Source of pain is a prior spinal fusion surgery
8. Has a cardiac pacemaker, implanted defibrillator or other implanted electronic device
9. Has radicular pain symptoms that affect functionality, quality of life or medication intake
10. Has undergone surgery to solve pain related to the study indication in the past 6 months
11. Patients with history of opioid, alcohol or drug abuse in the last 5 years, per investigator discretion
12. Any psychiatric condition that may interfere with the study assessments or prevent the subject from complying with the requirements of the protocol, in the judgement of the investigator
13. Inability to complete subjective data as required; e.g. on mobile application and questionnaires
14. Pregnant women (as determined by self-report)
15. Have severe epilepsy
16. Have severe form of cardiovascular disease
17. Any other disease, condition, or habit(s) that in the opinion of the Principal Investigator would interfere with study compliance or adversely affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walk Test | Once a week for 4 weeks
  Compare the change in patient's 6 Minute Walk Test (6MWT) between the Enso intervention group and the sham group using the validated 6MWT procedure.

SECONDARY OUTCOMES:
Functional back pain assessment | Once a week for 4 weeks
  Functional back pain assessment using a 0 to 10 Numeric Pain Intensity Scale, assessed immediately after the 6MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Tay, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No